CLINICAL TRIAL: NCT00685685
Title: A Single Dose Crossover Comparative Bioavailability Study of Lovastatin 40mg Tablets in Healthy Male Volunteers/Fasting State
Brief Title: Fasting Bioavailability Study of Lovastatin Tablets and Mevacor Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Kristin Arnold, Vice President R&D, Mutual Pharmaceutical Company
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: LVI-P4-125
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Therapeutic Equivalency
MeSH Terms: interventions — Lovastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lovastatin 40 mg tablet (Experimental): A single dose of Lovastatin 40 mg administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Lovastatin 40 mg tablets
- Lovastatin (Mevacor®) 40 mg Tablet (Experimental): A single dose of Lovastatin (Mevacor®) 40 mg administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Lovastatin (Mevacor®) 40 mg Tablets

INTERVENTIONS:
Drug: Lovastatin 40 mg tablets — 40 mg tablet administered after an overnight fast of at least 10 hours
  Arms: Lovastatin 40 mg tablet
Drug: Lovastatin (Mevacor®) 40 mg Tablets — 40 mg tablet administered after an overnight fast of at least 10 hours
  Other Names: Mevacor®
  Arms: Lovastatin (Mevacor®) 40 mg Tablet

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability and therefore the bioequivalence of a test formulation of lovastatin tablets to an equivalent dose of Mevacor® tablets after a single oral dose administered under fasting conditions.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability and therefore the bioequivalence of a test formulation of lovastatin tablets to an equivalent dose of Mevacor® tablets after a single oral dose administered under fasting conditions.

Fifty-four healthy, light/non/or ex-smoking, non-obese, male volunteers at least 18 years of age will be randomly assigned in a crossover fashion to receive each of two lovastatin dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, after an overnight fast of at least 10 hours, subjects will receive either a single oral dose of the test formulation, lovastatin (1 x 40 mg tablet), or a single oral dose of the reference formulation, Mevacor® (1 x 40 mg tablet). After a 7 day washout period on the morning of Day 8, following an overnight fast of at least 10 hours, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of lovastatin. Blood sampling will then continue on a non-confined basis at 36 and 48 hours post-dose. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drug and/or procedures. Vital signs will be monitored if judged necessary by the physician in charge. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Availability of volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form (ICF) duly signed by the volunteer
* Male aged of at least 18 with a body mass index (BMI) greater than or equal to 19 and below 30 kg/m²
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
* Healthy according to the laboratory results and physical examination
* Light, non- or ex-smokers. Light smokers are defined as someone smoking 10 cigarettes or less per day, and ex-smokers are defined as someone who completely stopped smoking for at least 3 months
* The informed consent form must be signed by all volunteers, prior to their participation in the study

Exclusion Criteria:

* Significant history of hypersensitivity to lovastatin or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability, including but not limited to cholecystectomy
* Presence of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of active liver disease or unexplained persistent elevations of serum transaminases
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of enzyme-modifying drugs in the previous 28 days before day 1 of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.)
* Participation in another clinical trial in the previous 28 days before day 1 of this study
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study
* Positive urine screening of drugs of abuse
* Positive results to HIV, HBsAg or anti-HCV tests

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-09; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Algorithme Pharma, Montreal, Canada

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Lovastatin 40 mg Tablets Then Mevacor® 40 mg Tablets: On the morning of Day 1 subjects received one tablet of the test formulation, Lovastatin 40 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received one tablet of the reference formulation, Mevacor® 40 mg, after an overnight fast of at least 10 hours.
- Mevacor® 40 mg Tablets Then Lovastatin 40 mg Tablets: On the morning of Day 1 subjects received one tablet of the reference formulation, Mevacor® 40 mg after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received one tablet of the test formulation, Lovastatin 40 mg, after an overnight fast of at least 10 hours.
Period: First Intervention
Arm/Group | Lovastatin 40 mg Tablets Then Mevacor® 40 mg Tablets | Mevacor® 40 mg Tablets Then Lovastatin 40 mg Tablets
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Lovastatin 40 mg Tablets Then Mevacor® 40 mg Tablets | Mevacor® 40 mg Tablets Then Lovastatin 40 mg Tablets
Started | 27 | 27
Completed | 25 | 26
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Lovastatin 40 mg Tablets Then Mevacor® 40 mg Tablets | Mevacor® 40 mg Tablets Then Lovastatin 40 mg Tablets
Started | 25 | 26
Completed | 25 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lovastatin 40 mg Tablets and Mevacor® 40 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either Lovastatin 40 mg or Mevacor® 40 mg following an overnight fast of at least 10 hours.
Arm/Group | Lovastatin 40 mg Tablets and Mevacor® 40 mg Tablets
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.5, 5, 5.5, 6, 7, 8, 10, 14, 18, 24, 36, and 48 hours after drug administration.
Population: Plasma concentration data for 51 of the 54 enrolled subjects were used in the statistical analysis. Two subjects were withdrawn from the study for adverse reactions and one subject withdrew his consent for personal reasons.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Lovastatin 40 mg Tablets; Mevacor® 40 mg Tablets: On the morning of Day 1 subjects received one tablet of either the test formulation, Lovastatin 40 mg, or the reference formulation, Mevacor® 40 mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received the alternate regimen following an overnight fast of at least 10 hours.
Arm/Group | Lovastatin 40 mg Tablets | Mevacor® 40 mg Tablets
Number analyzed (Participants) | 51 | 51
ng/mL | 1.86 (1.05) | 1.96 (1.02)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Lovastatin 40 mg Tablets | Mevacor® 40 mg Tablets
Number analyzed (Participants) | 51 | 51
ng-hr/mL | 30.64 (15.79) | 30.36 (17.28)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: 54 subjects were enrolled and 51 subjects completed the study. Lovastatin plasma concentration data for 48 subjects were used in the statistical analysis as the AUC(0-∞) was not calculated for 3 subjects. Mevacor® plasma concentration data for 50 subjects were used in the statistical analysis as the AUC(0-∞) was not calculated for 1 subject.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Lovastatin 40 mg Tablets | Mevacor® 40 mg Tablets
Number analyzed (Participants) | 48 | 50
ng-hr/mL | 34.52 (17.50) | 33.80 (18.97)

ADVERSE EVENTS:
Description: 54 subjects were enrolled in this study. Several subjects dropped out of the study prior to receiving both interventions. 53 subjects were administered lovastatin 40 mg tablest and 52 subjects were administered Mevacor® 40 mg tablets.
Groups:
- Lovastatin 40 mg Tablets; Mevacor® 40 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either Lovastatin 40 mg or Mevacor® 40 mg following an overnight fast of at least 10 hours.
Arm/Group | Lovastatin 40 mg Tablets | Mevacor® 40 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 10/53 | 7/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin 40 mg Tablets (N=53) | Mevacor® 40 mg Tablets (N=52)
loose stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
blood creatine phosphokinase increased (Investigations) | 2 (2) | 3 (3)
blood urea increased (Investigations) | 1 (1) | 1 (1)
heart rate decreased (Investigations) | 1 (1) | 0 (0)
neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 1 (1)
somnolence (Nervous system disorders) | 1 (1) | 0 (0)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
sweating increased (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pallor (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days